CLINICAL TRIAL: NCT01774799
Title: Educational Video to Improve Nursing Home Care in End-stage Dementia
Acronym: EVINCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Susan Mitchell, MD, Senior Scientist, Hebrew SeniorLife
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 12-013; R01AG043440 (NIH)
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Advanced Dementia
Keywords: advanced dementia; advance care planning; nursing home
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Advance care planning intervention (Experimental): At baseline, health care proxies in the intervention arm will be shown a 12-minute Advance Care planning video that describes 3 levels of treatment in advanced dementia: comfort basic and intensive. After viewing the video, the proxies will be asked their preferred level of care for the resident and this choice will be communicated to the residents primary care team in a written form.
  Interventions: Behavioral: Advance care planning intervention
- Usual care (Active Comparator): Residents in control nursing homes with receive the usual advance care planning that occurs in their nursing home.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Advance care planning intervention
  Arms: Advance care planning intervention
Other: Control group
  Arms: Usual care

SUMMARY:
This is a 5-year cluster RCT of a video Advance Care Planning intervention vs. control among 360 nursing home residents with advanced dementia (N=180/arm) in 20 matched nursing homes (10 intervention/10 control). Clinical outcomes will be collected at baseline, and quarterly (up to 12-months) regarding goals of care preferences, advance care planning, and treatments received. The primary outcome is decisions not to be hospitalized at 6 months.

DETAILED DESCRIPTION:
The over-riding goal of the EVINCE study is to conduct a cluster RCT of a video Advance Care Planning intervention in nursing home residents with advanced dementia. A total of 360 nursing home residents with advanced dementia (N=180/arm) in 20 matched nursing homes (10 intervention/10 control) will be recruited. These residents' proxies with also be recruited for a total sample size of 720 residents and proxies (resident/proxy dyads). Outcomes will be compared between residents in the intervention vs, control nursing homes at baseline and every 3 months up to 12 months. At baseline proxies of residents in the intervention nursing homes will view a 12-minutes video describing three level of care options in advanced dementia (intensive, basic and comfort) and their choice will be communicated to the resident's primary care providers. Residents in the control nursing homes will receive the usual advance care planning practiced in those facilities.

UPDATE SEPT 19, 2014: During the first 18 months of the study, recruitment of resident/proxy dyads was lower per facility than anticipated at the time of study design. Therefore, the number of matched pairs of NH recruited was increased. As of September 19, 2014, 19 NH pairs (38 NHs) were recruited and randomized with a plans to continue to up to 30 pairs as needed.

NHs were originally randomized using a paired approach matched for for-profit status and whether or not the NH had a special care dementia unit (SCU). In March 2014, the state of Massachusetts changed legislation defining an SCU. Many of the changes focused on specifics of staff training. As a result, SCUs in several participating facilities did not meet the new criteria and lost this official designation, although the actual clinical structure of the existing units did not change. Nonetheless, we opted to maintain the initial matching criteria of the first 19 NHs which included SCU based on the definition before the Massachusetts legislation change, but dropped this matching criterion after the legislation change. Thus, beginning with matched pair 20, NHs were matched solely on for-profit status.

UPDATE MARCH 2016 To reach subject recruitment numbers, additional facilities were recruited. As of this date, 60 NHs (30/arm) have been recruited, randomized and have had subject enrolled.

To achieve additional for power for Outcome 2, (aquisition of new decisions to forego hospitalizations) the target sample size was increased to 400.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65
* A diagnosis of dementia (any type)
* Global Deterioration Scale (GDS) score of 7
* Nursing home length of stay > 30 days
* Proxy is available who can speak in English
* Proxy must either live within a 60 mile radius of Boston or be available to come to the residents nursing home within 2 weeks of recruitment in order to conduct the in-person baseline interview.

Exclusion Criteria:

* Residents with cognitive impairment due to causes other than dementia (e.g. head trauma) and in short-term, sub-acute SNFs will be excluded

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 804 (Actual)
Dates: Start 2013-03; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Mitchell, MD, MPH, Principal Investigator — Hebrew SeniorLife; Angelo Volandes, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Hebrew Rehabilitation Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data form study are available through link porvided
Supporting Information: CSR
Time Frame: Now, indefinetly
Access Criteria: open
URL: https://ifar-dataverse.hsl.harvard.edu/dataverse/evince

REFERENCES:
- [Derived] Mitchell SL, Shaffer ML, Cohen S, Hanson LC, Habtemariam D, Volandes AE. An Advance Care Planning Video Decision Support Tool for Nursing Home Residents With Advanced Dementia: A Cluster Randomized Clinical Trial. JAMA Intern Med. 2018 Jul 1;178(7):961-969. doi: 10.1001/jamainternmed.2018.1506. PMID 29868778

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants are analyzed as dyads; proxies and patients.There are 402 dyads, for a total of 804 participants.
Groups:
- Advance Care Planning Intervention Residents: At baseline, health care proxies in the intervention arm will be shown a 12-minute Advance Care planning video that describes 3 levels of treatment in advanced dementia: comfort basic and intensive. After viewing the video, the proxies will be asked their preferred level of care for the resident and this choice will be communicated to the residents primary care team in a written form.
  Advance care planning intervention
- Usual Care (Control) Residents: Residents in control nursing homes with receive the usual advance care planning that occurs in their nursing home.
  Control group
- Advance Care Planning Intervention Proxies: At baseline, health care proxies in the intervention arm will be shown a 12-minute Advance Care planning video that describes 3 levels of treatment in advanced dementia: comfort basic and intensive. After viewing the video, the proxies will be asked their preferred level of care for the resident and this choice will be communicated to the residents primary care team in a written form.
- Usual Care (Control) Proxies: Proxies in control nursing homes experienced he usual advance care planning that occurs in their nursing home.
  Control group
Period: Overall Study
Arm/Group | Advance Care Planning Intervention Residents | Usual Care (Control) Residents | Advance Care Planning Intervention Proxies | Usual Care (Control) Proxies
Started | 212 | 190 | 212 | 190
Completed | 211 | 189 | 212 | 190
Not Completed | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Advance Care Planning Intervention Residents: Residents with advanced dementia in intervention group
- Usual Care (Control Group) Residents: Residents with advanced dementia in control group
- Advance Care Planning Intervention Proxies: Proxies of residents with advanced dementia in intervention group
- Usual Care (Control Group) Proxies: Proxies of residents with advanced dementia in control group
- Total: Total of all reporting groups
Arm/Group | Advance Care Planning Intervention Residents | Usual Care (Control Group) Residents | Advance Care Planning Intervention Proxies | Usual Care (Control Group) Proxies | Total
Number analyzed (Participants) | 212 | 190 | 212 | 190 | 804
Age, Continuous [Mean (Standard Deviation); unit: years] | 86.0 (7.4) | 87.4 (7.3) | 61.8 (10.9) | 62.8 (10.6) | 74.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 156 | 146 | 120 | 589
  Male | 45 | 34 | 66 | 70 | 215
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 178 | 172 | 177 | 173 | 700
  non-white | 34 | 18 | 35 | 17 | 104
Region of Enrollment [Number; unit: participants]
  United States | 212 | 190 | 212 | 190 | 804

OUTCOME MEASURES:

1. Primary Outcome: Documented Decisions to Forgo Hospitalization
Description: The proportion of residents with this outcome will be considered cumulatively at 6 months, including those who died; i.e., a composite of the percent of residents alive at six months who had a decision not to hospitalize and those who died before six months with this outcome prior to death. This cumulative outcome will only be based on time points following baseline as the baseline chart review data is conducted before the baseline proxy interview (i.e., before the proxy has seen the video in the intervention arm or heard options verbally in the control arm).
  (Decisions to forehospitalizations will be examined in a similar fashion at 3, 9, and 12 months, however the six month time frame is the primary trial outcome)
Time Frame: by six months
Measure: Count of Participants; unit: Participants
Groups:
- Advance Care Planning Intervention: At baseline, health care proxies in the intervention arm will be shown a 12-minute Advance Care planning video that describes 3 levels of treatment in advanced dementia: comfort basic and intensive. After viewing the video, the proxies will be asked their preferred level of care for the resident and this choice will be communicated to the residents primary care team in a written form.
  Advance care planning intervention
- Usual Care: Residents in control nursing homes with receive the usual advance care planning that occurs in their nursing home.
  Control group
Arm/Group | Advance Care Planning Intervention | Usual Care
Number analyzed (Participants) | 211 | 189
Participants | 133 | 119
Statistical Analysis 1: Comparison: Usual Care; Test type: Superiority; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.69 to 1.69]

2. Secondary Outcome: Acquisition of Decisions Not to Hospitalize
Description: This is a sub primary outcome. The modified ITT population will be the subgroup of residents who begin the study without a documented decision to forego hospitalization, and the outcome will be acquisition of a documented decision to forego hospitalization over the 12 month follow-up period. The analysis will utilize Cox proportional hazards regression. Results will be summarized using a hazard ratio and associated 95% confidence interval as well as plots of the cumulative incidence by group.
Time Frame: by 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Advance Care Planning Intervention | Usual Care
Number analyzed (Participants) | 108 | 92
Participants | 41 | 30
Statistical Analysis 1: Comparison: Advance Care Planning Intervention vs Usual Care; Test type: Superiority; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.66 to 2.20]

3. Secondary Outcome: Acquisition of Preference for Level of Care
Description: The proportion of proxies who have chosen comfort care (versus intermediate or intensive care) based on telephone interviews will be considered cumulatively at each assessment. At 6 months the outcome will include the proportion of proxies choosing comfort care up to and including the 6 month interview. Cumulative proportions will include data from the baseline interview for the control group, and baseline immediate post video interview for intervention group.The proportion of proxies choosing comfort care will be compared between the intervention and control groups using an extension of logistic regression based on general estimating equations (GEE) to account for clustering at the NH level at each time period.
Time Frame: 6 months
Population: Missing data are due to missing proxy interviews at certain follow-up time points
Measure: Count of Participants; unit: Participants
Arm/Group | Advance Care Planning Intervention | Usual Care
Number analyzed (Participants) | 209 | 182
Participants | 151 | 133
Statistical Analysis 1: Comparison: Advance Care Planning Intervention vs Usual Care; Test type: Superiority; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.58 to 1.58]

4. Other Pre Specified Outcome: Acquisition of Other Documented Advance Care Planning
Description: The proportion of residents who acquired a documented advance directive to forego tube-feeding will be compared in the intervention versus control group.
Time Frame: by 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Advance Care Planning Intervention | Usual Care
Number analyzed (Participants) | 211 | 189
Participants | 148 | 117
Statistical Analysis 1: Comparison: Advance Care Planning Intervention vs Usual Care; Test type: Superiority; Odds Ratio (OR) = 1.79, 95% CI 2-sided [1.13 to 2.82]

5. Other Pre Specified Outcome: Burdensome Treatments
Description: Burdensome treatments include: Hospitals transfers (hospitalizations or emergency room visits), tube feeding or parenteral therapy. The rate of burdensome treatments per 1000 resident days was compared between the intervention and control arms.
Time Frame: by 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Advance Care Planning Intervention | Usual Care
Number analyzed (Participants) | 211 | 189
Participants | 33 | 25
Statistical Analysis 1: Comparison: Advance Care Planning Intervention vs Usual Care; Test type: Superiority; p = 0.32, Regression, Linear

ADVERSE EVENTS:
Time Frame: 12 months
Description: The only adverse event that was monitored for was serious distress by proxy watching the video. The residents were NOT monitored for any adverse events
Groups:
- Advance Care Planning Intervention: Adverse events were only monitored in the health care proxies who viewed the video
  Advance care planning intervention
- Usual Care: Adverse event monitoring was no applicable the proxies in the usual care group as they did not watch the video, and the only adverse event monitored in the trial related to reactions to watching the video
  Control group
Arm/Group | Advance Care Planning Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 86/212 | 89/190
Serious Adverse Events (participants affected / at risk) | 0/212 | 0/0
Other Adverse Events (participants affected / at risk) | 0/212 | 0/190

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-12-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT01774799/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT01774799/SAP_001.pdf